CLINICAL TRIAL: NCT01242410
Title: Randomized Controlled Trial: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women With Short Cervix in Twins
Brief Title: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women With Short Cervix in Twins
Acronym: PECEP-TWINS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Responsible Party: Principal Investigator, Maria Goya, MD, PhD, PhD, Maternal-Infantil Vall d´Hebron Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pessary in twins TRIAL
Record Dates: First submitted 2010-09-28; First posted 2010-11-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-07

CONDITIONS: Preterm Birth
Keywords: Short cervix; Preterm birth; Cervical pessary; Twins
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expectant Management (No Intervention)
- Placement of cervical pessary since 23 weeks until 37 weeks (Experimental)
  Interventions: Device: Silicon ring (Arabin Cervical Pessary)

INTERVENTIONS:
Device: Silicon ring (Arabin Cervical Pessary) — Vaginal pessaries CE 0482 MED / CERT ISO 9003 /EN 46003
  Arms: Placement of cervical pessary since 23 weeks until 37 weeks

SUMMARY:
Placement of a vaginal pessary reduces significantly the rate of spontaneous preterm birth in pregnant women with twins and a short cervical length at 18-22 weeks scan.

DETAILED DESCRIPTION:
This trial includes pregnant women with twins undergoing routine ultrasound examination at 18.0 to 22.6 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Twins
* Minimal age of 18 years

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* Spontaneous rupture of membranes at the time of randomization
* Cervical cerclage in situ
* Active vaginal bleeding
* Placenta previa

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Spontaneous delivery before 34 completed weeks | Each 6 months

SECONDARY OUTCOMES:
Birth weight | Each 6 months
Fetal-Neonatal Death | Each 6 months
Neonatal morbidity | Each 6 months
Maternal adverse effects | Each 6 months
Preterm birth before 37 weeks or 28 weeks | Each 6 months
Rupture of membranes before 34 weeks | Each 6 months
Hospitalisation for threatened preterm labour | Each 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Carreras, Study Director — Hospital Vall d'Hebron; Maria M Goya, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Herbron, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Goya M, de la Calle M, Pratcorona L, Merced C, Rodo C, Munoz B, Juan M, Serrano A, Llurba E, Higueras T, Carreras E, Cabero L; PECEP-Twins Trial Group. Cervical pessary to prevent preterm birth in women with twin gestation and sonographic short cervix: a multicenter randomized controlled trial (PECEP-Twins). Am J Obstet Gynecol. 2016 Feb;214(2):145-152. doi: 10.1016/j.ajog.2015.11.012. Epub 2015 Nov 25. PMID 26627728